CLINICAL TRIAL: NCT01890655
Title: A Phase II, Multicentre Study to Evaluate the Long-term Safety and Efficacy of MT-1303 in Subjects With Relapsing-remitting Multiple Sclerosis Who Have Completed the MT-1303-E04 Study
Brief Title: Extension Study of MT-1303
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT-1303-E05
Record Dates: First submitted 2013-06-26; First posted 2013-07-02 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-04

CONDITIONS: Relapsing-remitting Multiple Sclerosis
Keywords: relapsing-remitting multiple sclerosis; RRMS
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- MT-1303-Low (Experimental): MT-1303-Low Dose
  Interventions: Drug: MT-1303-Low
- MT-1303-Middle (Experimental): MT-1303-Middle Dose
  Interventions: Drug: MT-1303-Middle
- MT-1303-High (Experimental): MT-1303-High Dose
  Interventions: Drug: MT-1303-High

INTERVENTIONS:
Drug: MT-1303-Low
  Arms: MT-1303-Low
Drug: MT-1303-Middle
  Arms: MT-1303-Middle
Drug: MT-1303-High
  Arms: MT-1303-High

SUMMARY:
To evaluate the long-term safety and tolerability of MT-1303 in subjects with relapsing remitting multiple sclerosis (RRMS).

ELIGIBILITY:
Inclusion Criteria:

* Completion of the 24-week treatment period in MT-1303-E04 as per protocol
* Able to provide written informed consent and to comply with the requirements of the protocol
* For males and females of reproductive potential, two methods of contraception must be used throughout the study and for 12 weeks after cessation of study medication. At least one of the methods of contraception must be a barrier method.

Exclusion Criteria:

* Permanent discontinuation of study medication prior to the end of treatment (EOT) visit in MT-1303-E04
* Newly diagnosed diabetes mellitus during MT-1303-E04

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 367 (Actual)
Dates: Start 2013-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Safety assessments | Month 18
  Adverse Events

SECONDARY OUTCOMES:
Clinical efficacy | Month 18
  Annualised relapse rate(ARR)
Magnetic Resonance Imaging (MRI) | Month 18
  Change and percent change in brain volume at EOT

CONTACTS AND LOCATIONS:
Overall Officials: Ludwig Kappos, MD, Study Director — University Hospital, Basel, Switzerland
Locations (17):
- Research Site, City Name, Belgium
- Research Site, City Name, Bulgaria
- Research Site, City Name, Canada
- Research Site, City Name, Croatia
- Research Site, City Name, Czechia
- Research Site, City Name, Finland
- Research Site, City Name, Germany
- Research Site, City Name, Hungary
- Research Site, City Name, Italy
- Research Site, City Name, Lithuania
- Research Site, City Name, Poland
- Research Site, City Name, Russia
- Research Site, City Name, Serbia
- Research Site, City Name, Spain
- Research Site, City Name, Turkey (Türkiye)
- Research Site, City Name, Ukraine
- Research Site, City Name, United Kingdom